CLINICAL TRIAL: NCT06727045
Title: The Effect of Mandala Art Therapy on Comfort Level in Patients Receiving Hemodialysis Treatment
Brief Title: The Effect of Mandala Art Therapy on Comfort Level in Patients Receiving HD Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Gül Kırıcı, Principal Investigator, Sanko University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SU-DON-GK-01
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Art Therapy; Mandala Painting; Hemodialysis Patients
Keywords: Hemodialysis; Nursing; Comfort; Mandala Painting

STUDY DESIGN:
Intervention Model Description: Groups (intervention-control) were determined by the minimization method by recording the scores obtained from age, gender and comfort performance.
Who Masked: Investigator
Masking Description: The minimization method was used to determine the patients in the intervention and control groups included in the research sample, and the random distribution of patients to the groups was made by a statistician other than the researcher using a computer program (www.randomizer.org) and taking into account age, gender, and scores from the comfort scale.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Questionnaire and Hemodialysis Comfort Scale Version-II (HDKS-II) were applied to the patients. Patients were randomised to groups. A literature review was conducted for the frequency and number of mandalas to be applied to the patients in the intervention group, and mandalas were applied during eight hemodialysis sessions every other day. Mandala painting was done approximately 30 minutes after the start of HD treatment, considering the art therapist's suggestion and the symptoms that may develop during HD. Each mandala painting was performed with a structured and different mandala pattern. In the study, a booklet called the "Mandala Booklet" consisting of eight structured mandala patterns with round shapes and containing general information about mandalas was used. The patients in the intervention group were informed face to face about the content of the booklet. At the end of the 17th day, the Hemodialysis Comfort Scale-Version II was applied to the group again.
  Interventions: Other: Mandala Coloring
- Control Group (No Intervention): Questionnaire and Hemodialysis Comfort Scale Version-II (HDKS-II) were applied to the patients. Randomization of the patients to the groups was done by a statistician other than the researcher with a computer program (www.randomizer.org) and was done by taking into account age, gender and comfort scale scores. No application was made to the patients in the control group. The booklet was given to the patients in the control group after the mandala coloring was completed. At the end of the 17th day, Hemodialysis Comfort Scale-Version II was applied to the group again.

INTERVENTIONS:
Other: Mandala Coloring — A literature review was conducted to determine the frequency and number of mandalas to be applied to the patients in the intervention group, and the average of the number of mandala sessions applied to different patient groups was obtained, and mandala application was performed during a total of eight hemodialysis sessions, every other day. Mandala painting was performed approximately 30 minutes after the start of HD treatment, considering the art therapist's recommendation and the symptoms that may develop during HD. Each mandala painting was performed with a structured and different mandala pattern. Since it was stated that the use of round patterns instead of square patterns was effective in increasing the comfort level, the booklet called "Mandala Booklet", consisting of 8 structured mandala patterns with round shapes and containing general information about mandala, was used in the study. The group was informed about the content of the booklet face to face. Dry pencils were prefer
  Arms: Intervention Group

SUMMARY:
This study was conducted to evaluate the effect of mandala painting on the comfort level of patients receiving HD treatment.

DETAILED DESCRIPTION:
The number of patients diagnosed with end-stage renal disease (ESRD) is constantly increasing and the most common method used in the treatment of these patients is hemodialysis (HD). HD is the process of passing the blood taken from the patient through the HD device, regulating fluid and electrolytes, and cleaning waste products such as urea. The aim of this process is to prevent complications, strengthen self-care, and thus increase the patient's quality of life and ensure their comfort. However, patients who receive HD treatment have to deal with various problems. This situation negatively affects the comfort of the HD patient. In addition, many factors such as constantly going to a dialysis center for the HD procedure, restriction of movements during the HD session, and disruption of work harmony and social relationships reduce the comfort of the patients. Therefore, ensuring the comfort of the HD patient is very important. A number of integrative methods are recommended to increase comfort. One of these methods, mandala, is effectively used in the field of art therapy. Mandala, which has a long history and represents integrity, is a Sanskrit word that means "circle" or completion and increases the individual's personal awareness. According to art psychotherapists, mandala painting is one of the main tools of other art psychotherapy techniques that focus on healing. Mindfulness-based activities such as drawing or painting mandalas allow the person to keep their attention in the "moment", make sense of what they have MINIMIDAted, increase their well-being and feel more comfortable. Mandala, which is a concentration method, helps the person stay in the moment. Energy and emotions can also change with the effects of the colors used. It is also emphasized that mandala painting contributes to symptom management, can be used in all age groups and has a positive effect on the treatment process of different diseases and disorders. The natural calming effect of mandala on the mind and body not only strengthens the desire to heal, but also helps the person get rid of psychological fragmentation. In line with these data, it is thought that activities such as mandala can be effective in HD patients who are faced with a large number of stress factors. Therefore, the effect of mandala painting on the comfort level of patients receiving HD treatment was evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18-65
* Those with no communication problems
* Those who can understand and speak Turkish
* Those who have been receiving HD treatment for at least three months
* Those who have been receiving HD three times a week
* Those who have no visual impairment
* Those who do not have any problems affecting fine motor function in the upper extremities (such as rheumatoid arthritis)
* Those who volunteered to participate in the study were included in the study

Exclusion Criteria:

* Patients with arteriovenous fistula in the dominant arm
* Patients who had previously undergone mandala application were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2023-12-29 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Hemodialysis Comfort Scale Version-II | At the beginning and at the end of the 17th day
  Due to the insufficient number of items in the previously developed Hemodialysis Comfort Scale, Koşar and colleagues developed the Hemodialysis Comfort Scale-Version II (HDKÖ-II) scale and its validity and reliability study was conducted by the same authors. The scale consists of 26 items and the responses to the items were prepared in a five-point Likert type as never, very rarely, sometimes, very often, always. The scale has six sub-dimensions as physical relief, physical relaxation, psychospiritual relaxation, psychospiritual empowerment, environmental empowerment, and sociocultural relaxation. Although there are reverse and direct scored items in the scale, the number of reverse scored items is high. As the score obtained from the scale increases, the patient's comfort also increases.

SECONDARY OUTCOMES:
Question Form | At the beginning
  The questionnaire form was created by the researchers in line with the literature. Questions 1-11 of this form include a total of 21 questions, questioning the descriptive characteristics of the patients, questions 12-21 questioning the HD treatment and the emotions felt by the patients during the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Nimet Ovayolu, Prof. Dr., Study Director — Sanko University
Locations (1):
- Private Damla dialysis center, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No